CLINICAL TRIAL: NCT03477929
Title: Cetrorelix and Ganirelix Flexible Protocol for In Vitro Fertilization: a Prospective Randomized Trial
Brief Title: Cetrorelix and Ganirelix Flexible Protocol for (IVF)
Acronym: IVF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi 'G. d'Annunzio' Chieti e Pescara (Other)
Responsible Party: Principal Investigator, Antonia Iacovelli, Principal Investigator, Università degli Studi 'G. d'Annunzio' Chieti e Pescara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cetrorelix-Ganirelix
Record Dates: First submitted 2018-02-28; First posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Infertility/Sterility
Keywords: In vitro fertilization; gnrh antagonist; pituitary suppression
MeSH Terms: conditions — Infertility | interventions — ganirelix; cetrorelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ganirelix (Experimental): multiple dose of Ganirelix acetate (0.25mg) are administered when the lead follicle is ≥ 14 mm until hCG criteria are met
  Interventions: Drug: Ganirelix Acetate
- cetrorelix (Experimental): multiple dose of Cetrorelix acetate (0.25mg) are administered when the lead follicle is ≥ 14 mm until hCG criteria are met
  Interventions: Drug: Cetrorelix Acetate

INTERVENTIONS:
Drug: Ganirelix Acetate — multiple dose of Ganirelix acetate (0.25mg) are administered when the lead follicle is ≥ 14 mm until hCG criteria are met
  Arms: ganirelix
Drug: Cetrorelix Acetate — multiple dose of Cetrorelix acetate (0.25mg) are administered when the lead follicle is ≥ 14 mm until hCG criteria are met
  Arms: cetrorelix

SUMMARY:
Recombinant gonadotropins are currently used for ovarian stimulation in women undergoing to IVF for infertility. Recently new flexible protocols have been introduced: the "single dose" and "multiple dose" protocol. The single dose protocol is performed just using Cetrorelix by the administration of a single injection of Cetrorelix 3 mg subcutaneous when the lead follicle is ≥ 14 mm. The multiple dose protocol consider the daily administration of Cetrorelix 0.25 mg subcutaneous or Ganirelix 0.25 mg subcutaneous when the lead follicle is ≥ 14 mm and until the realization of hCG criteriaThere are few data from letterature about the comparison of the efficacy in pitituary suppression and pregnancy outcome of Ganirelix and Cetrorelix.

Objective: to compare the efficacy in pituitary gonadotropin suppression and IVF outcome of multiple dose flexible gonadotrophin-releasing hormone (GnRH) antagonist administration according to follicular size using daily injection of Cetrorelix or Ganirelix.

Interventions : patients are randomly assigned in to Cetrorelix acetate group or Ganirelix acetate group. Multiple dose of Cetrorelix acetate (0.25 mg) or multiple dose of Ganirelix acetate (0.25mg) are administered when the lead follicle is ≥ 14 mm until hCG criteria are met.Oocyte maturation trigger is performed by the administration of subcutaneous r-hCG (250 μg) or of intramuscular hCG (10,000 IU). After 36 hour transvaginal oocyte retrieval is performed followed by ICSI and embrio transfer (72 hours later).

ELIGIBILITY:
Inclusion criteria :

* 18-39 hyears old with regular menstrual cycles (25-35 days in length);
* Body Mass Index between 18-29 kg\m2
* Basal follicle-stimulating hormone levels within normal range (<30 mUI\mL)
* Absence of clinically relevant anomalies at transvaginal ultrasound examinatio

Exclusion Criteria:

* Patients affected by grade III or IV endometriosis according to American Society for Reproductive Medicine (ASRM)
* History of Ovarian Hyperstimulation Stimulation (OHSS)
* History of poor response in previous IVF\ICSI cycle: ≤ 3 oocytes retrieved
* ≥ 3 prior consecutive IVF\ICSI cycle without a clinical pregnancy.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-12-15 (Estimated); Study Completion 2019-01-15 (Estimated)

PRIMARY OUTCOMES:
serum LH levels | through study completion,an average of 9 months
  percentage of patients not having serum levels of LH ≥ 10IU\L (defined as premature LH surge) on the day of hCG administration.

SECONDARY OUTCOMES:
number of follicles ≥ 14mm on the day of hCG administration | through study completion,an average of 9 months
  number of follicles ≥ 14mm
FSH serum levels on the day of hCG administration | through study completion,an average of 9 months
  mUI/ml
FSH on the day of antagonist administration | through study completion,an average of 9 months
  mUI/ml
FSH serum level on the day after the antagonist administration | through study completion,an average of 9 months
  mUI/ml
LH serum level on the day of antagonist administration | through study completion,an average of 9 months
  mUI/ml
LH serum level on the day after the antagonist administration | through study completion,an average of 9 months
  mUI/ml
E2 serum level on the day of antagonist administration | through study completion,an average of 9 months
  mUI/ml
E2 serum level on the day after the antagonist administration | through study completion,an average of 9 months
  mUI/ml
number of oocyte retrieved | through study completion,an average of 9 months
  how many oocyte were retrieved on transvaginal oocyte retrieval
number of metaphase II oocyte retrieved | through study completion,an average of 9 months
  how many metaphase II oocyte were retrieved on transvaginal oocyte retrieval
embryos obtained for patients | 72 hours after transvaginal oocyte retrieval
  how many embryos were obtained for patient for each arm
grade A embryos transferred | 72 hours after transvaginal oocyte retrieval
  number of grade A embryo were transferred for patient
total dose of gonadotropins administered | through study completion,an average of 9 months
  number of Units of gonadotropin administered for Controlled Ovarian Hyperstimulation
duration of gonadotropin treatment | through study completion,an average of 9 months
  how many days were necessary to complete the Controlled Ovarian Hyperstimulation
percentage of patients developing OHSS | 15 days after the transvaginal oocyte retrieval
  how many patient for each arm develop OHSS (Ovarian Hyperstimulation Syndrome)
implantation rate | 30 days after the embyo transfer
  The number of gestational sacs observed divided by the number of embryos transferred.
pregnancy rate | 14 days after the transvaginal oocyte retrieval
  The number of clinical pregnancy (Positive hCG test) divided by the number of embryos transferred

CONTACTS AND LOCATIONS:
Overall Officials: Gian Mario Tiboni, professor, Study Director — Università degli Studi 'G. d'Annunzio' Chieti e Pescara
Locations (1):
- Ospedale Bernabeo, Ortona, Chieti, Italy

IPD SHARING:
Plan to Share IPD: No